CLINICAL TRIAL: NCT03812536
Title: Spontaneous Void Requirements for Patients Undergoing Ambulatory Anorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syed Husain (Other)
Responsible Party: Sponsor-Investigator, Syed Husain, Assistant Professor - Colon and Rectal Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0208
Record Dates: First submitted 2018-05-24; First posted 2019-01-23 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Complications, Postoperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC Voiding Protocol (No Intervention): Patients in the control group will follow the standard of care protocol and are required to void post anorectal surgery before being discharged home.
- No Void Intervention (Experimental): Patients in the experimental group (No Void Intervention) will be discharged home without voiding spontaneously.
  Interventions: Other: No Void

INTERVENTIONS:
Other: No Void — Currently the protocol at The Ohio State University Hospital requires voiding spontaneously prior to discharge from the PACU. Our intervention group will be discharged home without having to void spontaneously as a discharge criteria.
  Arms: No Void Intervention

SUMMARY:
The objective of this study is to assess if not requiring patients to spontaneous void prior to discharge from the post-anesthesia care unit (PACU) will results in shorter lengths of stay in the post-anesthesia care unit without increasing hospital readmissions or emergency room visits.

DETAILED DESCRIPTION:
This study will be a prospective clinical trial, in which 100 anorectal surgery patients will be randomly assigned to a control (spontaneous void) or experimental (no void group). The spontaneous void group will include 50 patients who will be required to void spontaneously after anorectal surgeries. The no void group will be 50 patients who will be discharged home from the PACU once they meet ambulatory surgery center discharge criteria per hospital guidelines. Patients requiring anorectal surgeries will be consented to take part in the study during the preoperative outpatient office visit. A post-operative phone call will be made by designated study personnel to participants on post-op day 30 using a study questionnaire to assess re-admission and emergency room visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Patients undergoing hemorrhoidectomy, fistulotomy or anal condyloma excision

Exclusion Criteria:

* Age < 18 yo or > 80 yo
* Prisoners
* Pregnant Women
* Unable or unwilling to follow the study protocol or any reason the research team believes the subject is not appropriate candidate for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Husain, MBBS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC Voiding Protocol | No Void Intervention
Started | 47 | 57
Completed | 44 | 56
Not Completed | 3 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients undergoing ambulatory surgeries for 1. Hemorrhoids, 2. Anal fistula and 3. Anal Condyloma.
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC Voiding Protocol | No Void Intervention | Total
Number analyzed (Participants) | 44 | 56 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 53 | 94
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 42 [24 to 72] | 41 [18 to 71] | 42 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 26 | 39 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 41 | 77
  African American | 5 | 12 | 17
  Asian | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 44 | 56 | 100
Disease Condition 1. Hemorrhoids. 2. Fistula. 3. Anal Condyloma 4. Exam Under Anesthesia [Count of Participants; unit: Participants]
  Hemorrhoidectomy | 7 | 6 | 13
  Fistulotomy | 10 | 19 | 29
  Exam Under Anesthesia | 14 | 16 | 30
  Condyloma | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: PACU Time
Description: This is the time patients in each arm spend in recovery. Measured as minutes elapsed between the end of surgery (surgery end time) and discharge from recovery room.
Time Frame: This measure will be recorded through the study period.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | SOC Voiding Protocol | No Void Intervention
Number analyzed (Participants) | 44 | 56
Minutes | 129.1 (100.0) | 210.0 (175.0)

2. Secondary Outcome: 30-day Readmission
Description: Number of patients readmitted in the 30-days period after surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- SOC Voiding Protocol: Patients in the control group will follow the standard of care protocol and are required to void post anorectal surgery before being discharged home.
  No 30-day readmissions were noted.
- No Void Intervention: Patients in the experimental group (No Void Intervention) will be discharged home without voiding spontaneously.
  No Void: Currently the protocol at The Ohio State University Hospital requires voiding spontaneously prior to discharge from the PACU. Our intervention group will be discharged home without having to void spontaneously as a discharge criteria.
  No 30-day readmissions were noted.
Arm/Group | SOC Voiding Protocol | No Void Intervention
Number analyzed (Participants) | 44 | 56
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days.
Arm/Group | SOC Voiding Protocol | No Void Intervention
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/56
Other Adverse Events (participants affected / at risk) | 0/44 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03812536/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03812536/ICF_001.pdf